CLINICAL TRIAL: NCT02447653
Title: A Randomised Controlled Study Comparing Hydroxyapatite (HA) Coating Versus Plasma Porous Spray in Press-fit Acetabular Components Early Outcomes With Dual Energy X-ray Absorptiometry (DEXA)
Brief Title: Hydroxyapatite (HA) Coating Versus Plasma Porous Spray (PPS) in Press-fit Acetabular Components Early Outcomes With DEXA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMETAU09
Record Dates: First submitted 2015-05-08; First posted 2015-05-19 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydroxyapatite Coating (Experimental): G7 HA Acetabular component will be implanted
  Interventions: Device: G7 HA Acetabular Component
- Plasma Porous Spray (Active Comparator): G7 PPS Acetabular component will be implanted
  Interventions: Device: G7 PPS Acetabular Component

INTERVENTIONS:
Device: G7 HA Acetabular Component — G7 HA Acetabular Component
  Arms: Hydroxyapatite Coating
Device: G7 PPS Acetabular Component — G7 PPS Acetabular Component
  Arms: Plasma Porous Spray

SUMMARY:
The study design comprises a randomized trial of patients undergoing primary total hip arthroplasty using the G7 acetabular system and Taperloc Complete stem comparing regular plasma porous spray with HA coating using Bonemaster (BM) in an uncemented cup. DEXA scanning will be used to measure periprosthetic bone mineral density. Clinical evaluations will be conducted .

DETAILED DESCRIPTION:
The study design comprises a randomized trial of patients undergoing primary total hip arthroplasty using the G7 acetabular system and Taperloc Complete stem comparing regular plasma porous spray with HA coating using Bonemaster (BM) in an uncemented cup. DEXA scanning will be used to measure periprosthetic bone mineral density preoperatively and post-operatively at 6 weeks, 12 weeks, 26 weeks, and 12 months for both the treated and contralateral hip joint. Clinical evaluations will be conducted preoperatively, and postoperatively at 6, 12, 26 weeks, 12 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with osteoarthritis who are candidates for a primary total hip replacement with uncemented acetabular and femoral components as determined by the surgeon.
2. Male and non-pregnant female patient aged 18 to 70.
3. Patients who understand the conditions of the study and are willing to participate for the length of the prescribed follow-up.

Exclusion Criteria:

1. Patients requiring total hip replacement surgery for a fresh hip fracture.
2. Patients with inflammatory arthritis
3. Patients with metabolic bone disease or taking drugs that affect bone turnover. 4 .Patients requiring revision surgery of a previously implanted total hip replacement system or patients requiring a conversion surgery from a previous fracture fixation or hip fusion.

5. Patients with presence of malignancy in the area of the involved hip joint. 6. Patients who, as judged by the surgeon, are mentally incompetent or are reasonably unlikely to be compliant with the prescribed postoperative routine and the follow-up evaluation schedule.

7. Patients with other concurrent illnesses that are likely to affect their outcome such as sickle cell anaemia, systemic lupus erythematosus or renal disease requiring dialysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Bone Remodelling (DEXA analysis) | 12 months
  DEXA analysis

SECONDARY OUTCOMES:
Clinical (Harris Hip Score) | 24 months
  Harris Hip Score
Clinical (Oxford Hip Score) | 24 months
  Oxford Hip Score

CONTACTS AND LOCATIONS:
Overall Officials: David Liu, Principal Investigator — Gold Coast Centre for Bone and Joint Surgery
Locations (1):
- Greenslopes Private Hospital, Greenslopes, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No